CLINICAL TRIAL: NCT03296189
Title: Intraluminal Ureteric Injection of High Concentration Alkalinised Long-acting Local Anaesthetic and STeroid Post urEteroscopy: A Prospective Double Blinded Randomised Controlled Trial (LASTE Trial)
Brief Title: Local Anaesthetic and Steroid in the Ureter
Acronym: LASTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Adelaide and Meath Hospital, incorporating The National Children's Hospital (Other)
Responsible Party: Principal Investigator, Rustom P Manecksha, MD, FRCS (Urol.), Principal investigator, The Adelaide and Meath Hospital, incorporating The National Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AMNCH-GU-2017-2
Record Dates: First submitted 2017-09-08; First posted 2017-09-28 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Pain, Postoperative; Ureter Stone
Keywords: ureteroscopy; ureteric stent; intraluminal; local anaesthetic/anesthetic; steroid/glucocorticoid
MeSH Terms: conditions — Pain, Postoperative; Ureterolithiasis | interventions — Levobupivacaine; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: Three arm double-blinded prospective randomised controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: 10 mls of solution will be handed to operating surgeon by the scrub nurse. The nurse will be the only person aware of the solution content and it will be documented discreetly. The operating surgeon, the investigator and the patients will not be aware of the solution used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local anaesthetic (Active Comparator): Post-ureteroscopy intraluminal injection of alkalinised high concentration levo-bupivicaine in the renal pelvis
  Interventions: Drug: Levobupivacaine
- Local anaesthetic + steroid (Active Comparator): Post-ureteroscopy intraluminal injection of 10 mls alkalinised high concentration levo-bupivicaine with l dexamethasone in the renal pelvis
  Interventions: Drug: Dexamethasone Sodium Phosphate
- Placebo (Placebo Comparator): Post-ureteroscopy intraluminal injection of 10 mls normal saline (placebo) in the renal pelvis
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Levobupivacaine — intraluminal injection post procedure for pain relief: alkalinised high concentration 10 mls
  Arms: Local anaesthetic
Drug: Dexamethasone Sodium Phosphate — intraluminal injection post procedure for pain relief: alkalinised high concentration 10 mls levobupivicaine and 2mls dexamethasone
  Arms: Local anaesthetic + steroid
Drug: Placebos — 10 mls normal saline
  Arms: Placebo

SUMMARY:
Précis:

Randomised control trial to evaluate safety and efficacy of intraluminal injection of high pH-high concentration of a long-acting local anesthetic and long-acting glucocorticoid in the ureter after ureteroscopy.

Objectives:

To evaluate a novel method to ameliorate post-ureteroscopy pain in all patients (with and without stents)

Endpoints:

Primary endpoint: mean visual analog pain scale (VAS) post-operatively starting at 1 hour, 4 hours, 8 hours, 24 hours and 7 days post-procedure (minimum of 3 VAS scores). VAS pain, ureteral stent symptoms and analgesic requirement will be assessed at different points during this time period.

Secondary endpoint: Postoperative Nausea/Vomiting (PONV), safety of intraluminal injection of high concentration alkalinized local anaesthetic solution by comparing adverse events between placebo and treatment arms. In addition, rehospitalisation rates and postoperative length of stay will be compared between the three groups.

Population:

150 adult patients undergoing ureteroscopy for ureteric stone disease stratified into negative ureteroscopy and those treated for a stone with or without stent insertion postoperatively Number of Sites: Tallaght Hospital Study Duration: 8 months

DETAILED DESCRIPTION:
Study Rationale Ureteroscopy is a widely performed procedure in urology. Pain is one of the commonest complications after ureteroscopy and one of the common reasons for re-admission after this procedure. Insertion of a stent post-ureteroscopy can cause pain affecting daily activities in 80% of the patients. Pain post ureteroscopy is multi-factorial and currently there is no specific method used clinically to treat this. Intraluminal injection of local anesthetic solution in the ureter has been extensively studied in the animal model with positive results. Intraluminal injection steroids has also been studied previously and steroids have also been used in medical expulsive therapy for ureteric stones previously. The investigators are proposing the use of high concentration alkalinized long-acting local anaesthetic levo-bupivicaine and long-acting steroid dexamethasone for post-ureteroscopy pain. It is simple, cheap, safe, easy to perform and widely available.

Background Intraluminal injection of local anesthetics (LA) in the ureter has been studied previously in animal models. Burdgya et al in 1986, USSR examined effects of LA on guinea pig ureters . Action potential of ureteric smooth muscle has initial fast component consisting of repeated gradually decaying spikes and a subsequent slow component i.e plateau. This action potential is accompanied by a brief contraction. Two opposite effects of LA occur on ureteric smooth muscle: Low concentrations of procaine, lignocaine and tetracaine (0.1-1 mM) at pH 7.4 increased duration of slow plateau of the evoked action potentials. At higher concentrations lignocaine (5mM) and tetracaine (0.5mM) caused complete inhibition of evoked action potentials and phasic contractions. Procaine 5mM predominantly inhibited contractile responses. High pH (9) significantly increased while low pH (pH 6) decreased the inhibitory action of procaine and lignocaine. Tetracaine had the most potent inhibitory action on ureter smooth muscle with the weakest stimulant action while lignocaine had stronger inhibitory effect on ureter smooth muscle than procaine. Ross et al in 1972 reported intraluminal injection of 2% lignocaine reduced peristaltic activity in 5 out of 15 ureters in their patients with no effect in the remaining group.

Andersson and Ulmsten found that local instillation of 4% lignocaine in their patients caused an initial brief stimulation followed by reduced activity. Tsuchida in 197 studied dog ureters to report prompt inhibitory effect of 4% lignocaine applied to mucosa invivo with no effect when applied to adventitia.

Struthers in 1976 in his invivo dog studies found both systemic and intraluminal administration of lignocaine, procaine and mepivacaine caused only hyperperistalsis and never inhibition. Sur et al published a study with intravesical injection of ropivacaine before ureteroscopic surgery demonstrated trends toward decreased pain and voiding symptoms. Patients received five injections of 2 mL 0.5% ropivacaine around the ureteral orifice or to the control cohort, who received five injections of 2 mL of 0.9% normal saline in identical locations. A pilot study suggested that PSD597 (intravesical alkalinized lidocaine) is effective for treating interstitial cystitis/painful bladder syndrome (IC/PBlS) , providing short-term amelioration of symptoms in a substantial proportion of patients, with a strong suggestion that repeating the treatment has a potentially cumulative effect. A randomized controlled trial comparing injection of non-irritating salt water (placebo), and half an injection of pH buffered lidocaine before the stent placement in patients undergoing ureteroscopy is currently being conducted. Till date there is no human study assessing the efficacy and safety of high concentration alkalinised long-acting LA injection for post-ureteroscopy pain based on the results of the animal studies outlined above.

The anaesthetic drug chosen for this study is levobupivacaine (Chirocaine™ -): it is S-isomer of bupivacaine, an amino-amide local anaesthetic widely used in regional anaesthesia, in postoperative analgesia and in treatment of acute and chronic pain. This drug produces sensory and motor nerve conduction block, acting on sodium channels of the cell membrane - sensitive to electric stimulus - but also on potassium and calcium channels. Moreover, it is remarkable for a rapid onset time and a long duration. In vitro and in vivo pharmacodynamic studies show that levobupivacaine has the same potency as bupivacaine, though the former is less likely to cause cardio- and neurotoxicity.

The effect of steroids on ureteric motility has previously been studied in in-vitro sheep models. Glucocorticoids inhibit the release of phospholipase A2 enzyme which catalyses the release of arachidonic acid from membrane phospholipids and thereby can have a spasmolytic action on the ureter by a prostaglandin-inhibitory action. Dexamethasone has shown the most potent dose dependant effect on the ureteral motility, it blocks ureteral motility in high concentrations within 24 minutes of instillation. Being a long-acting steroid, its duration of action in previous studies on nerve blocks and intra-articular injections is demonstrated at 12 weeks.

Study population: 150 patients undergoing ureteroscopy for ureteric stones:

1. Ureteric stone treatment (including proximal, mid and distal ureteric stones) with or without JJ stent insertion OR
2. Negative ureteroscopy (no stone found)

Pre and intraop: Obtain informed written consent pre-operatively with a pre-operative pain score, and rule out any allergies. Standardised uniform anesthetic regimen in all ureteroscopies.Post-ureteroscopy: drain the renal pelvis

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing ureteroscopy for ureteric stone disease
* Able to undergo a general anaesthetic
* At least 18 years old
* Willing and able to complete patient symptom questionnaires

Exclusion Criteria:

* Solitary Kidney
* Renal failure
* Anatomic bladder or ureteral abnormality
* Uncorrected coagulopathy
* Previous cystectomy or urinary diversion
* Neurogenic bladder
* Interstitial cystitis
* Transplanted kidney
* Pregnancy
* Requires an indwelling catheter
* Recurrent urinary tract infections
* Pelvic kidney
* Requires bilateral treatment/stents
* Previous bladder or ureteral reconstructive surgery
* Ureteral perforation during procedure
* Known sensitivity to lidocaine
* Febrile at time of randomization or treatment
* Requires spinal anaesthetic
* Stenting without stone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain | at up to 7 days post op
  Visual Analog Pain Scale (VAS) at least 3 different time points post-ureteroscopy

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) | at up to 7 days post op
Length of stay post-op | at up to 7 days post op
rehospitalisation rate | at up to 7 days post op
Need for analgesia | at up to 7 days post op

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaide and Meath incorporating National Children's hopsital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El Harrech Y, Abakka N, El Anzaoui J, Ghoundale O, Touiti D. Ureteral stenting after uncomplicated ureteroscopy for distal ureteral stones: a randomized, controlled trial. Minim Invasive Surg. 2014;2014:892890. doi: 10.1155/2014/892890. Epub 2014 Nov 9. PMID 25431663
- [Background] Burdyga ThV, Magura IS. The effects of local anaesthetics on the electrical and mechanical activity of the guinea-pig ureter. Br J Pharmacol. 1986 Jul;88(3):523-30. doi: 10.1111/j.1476-5381.1986.tb10232.x. PMID 3742148
- [Background] Ross JA EP, Kirkland IS. Ibid. 1972:125.
- [Background] Andersson KE, Ulmsten U. Effects of spinal anaesthesia, lidocaine, and morphine, on the motility of the human ureter in vivo. Scand J Urol Nephrol. 1975;9(3):236-42. doi: 10.3109/00365597509134219. PMID 1209180
- [Background] Boyarsky ASaS. The Pharmacology of the Urinary Tract. In: Caine M, editor.1984.
- [Background] Sur RL, Haleblian GE, Cantor DA, Springhart WP, Albala DM, Preminger GM. Efficacy of intravesical ropivacaine injection on urinary symptoms following ureteral stenting: a randomized, controlled study. J Endourol. 2008 Mar;22(3):473-8. doi: 10.1089/end.2007.9847. PMID 18290733
- [Background] Nickel JC, Moldwin R, Lee S, Davis EL, Henry RA, Wyllie MG. Intravesical alkalinized lidocaine (PSD597) offers sustained relief from symptoms of interstitial cystitis and painful bladder syndrome. BJU Int. 2009 Apr;103(7):910-8. doi: 10.1111/j.1464-410X.2008.08162.x. Epub 2008 Nov 13. PMID 19021619
- [Background] The American Heritage® Stedman's Medical Dictionary. http://www.dictionary.com/browse/life-expectancy. Accessed 13/12/16. 2002.
- [Background] Angelo-Khattar M, Thulesius O, Cherian T. The effect of glucocorticosteroids on in vitro motility of the ureter of the sheep. Br J Pharmacol. 1989 Mar;96(3):527-30. doi: 10.1111/j.1476-5381.1989.tb11849.x. PMID 2720291
- [Background] Manchikanti L, Manchikanti KN, Manchukonda R, Cash KA, Damron KS, Pampati V, McManus CD. Evaluation of lumbar facet joint nerve blocks in the management of chronic low back pain: preliminary report of a randomized, double-blind controlled trial: clinical trial NCT00355914. Pain Physician. 2007 May;10(3):425-40. PMID 17525777